CLINICAL TRIAL: NCT03237572
Title: Focused Ultrasound Therapy to Augment Antigen Presentation and Immune-Specificity of Checkpoint Inhibitor Therapy With Pembrolizumab in Metastatic Breast Cancer
Brief Title: Focused Ultrasound and Pembrolizumab in Metastatic Breast Cancer
Acronym: Breast-48
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low rate of enrollment
Sponsor: Patrick Dillon, MD (Other)
Responsible Party: Sponsor-Investigator, Patrick Dillon, MD, Associate Professor, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19900
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Results first posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; pembrolizumab; focused ultrasound; immunotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Pilot, 2-arm randomized study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Arm A: 1st dose of pembrolizumab after HIFU (Experimental): Pembrolizumab (200 mg) administered intravenously, days 22, 43, 64, followed by day 1 of each ensuing 3 -week cycle. Focused ultrasound tumor ablation day 15. High-intensity focused ultrasound ablation will target 50% of the tumor, up to 3 cubic centimeters.
  Interventions: Drug: Pembrolizumab; Device: High-intensity focused ultrasound (HIFU)
- Arm B: 1st dose of pembrolizumab before HIFU (Experimental): Pembrolizumab (200 mg) intravenously, days 1, 22, 43, 64, followed by day 1 of each ensuing 3 -week cycle. Focused ultrasound tumor ablation day 15. High-intensity focused ultrasound ablation will target 50% of the tumor, up to 3 cubic centimeters.
  Interventions: Drug: Pembrolizumab; Device: High-intensity focused ultrasound (HIFU)

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab (200 mg)
  Other Names: Keytruda
Device: High-intensity focused ultrasound (HIFU) — Ablation will target 50% of the tumor, up to 3 cubic centimeters

SUMMARY:
This pilot study evaluates the use of high-intensity focused ultrasound (HIFU) combined with pembrolizumab in patients with metastatic breast cancer. One-half of participants will be randomized to receive the first dose of pembrolizumab after HIFU and one-half of participants will be randomized to receive their first dose of pembrolizumab before HIFU.

ELIGIBILITY:
Inclusion Criteria (summary):

* Histologically confirmed metastatic or unresectable breast cancer
* Any receptor status (estrogen receptor, progesterone receptor, HER2 receptor). Patients who are HR+ should also no longer be candidates for hormonal-based therapy. Patients who are HER2+ should have progressed on or no longer be candidates for available HER2 directed therapy. Hormonal therapy must be stopped prior to day 1 of treatment.
* Patients must have had at least one prior line of therapy for breast cancer in the metastatic setting.
* Patients must have an accessible lesion in the breast/chest wall/axilla which has not been previously thermally ablated. Prior breast irradiation is acceptable if the lesion has recurred or grown following radiation.
* Patients must agree to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication.
* Patients must have at least one target lesion in breast/chest wall/axilla which is amenable to application of high intensity focused ultrasound:
* Patients must be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion.
* Performance status of 0 or 1 on the ECOG Performance Scale.
* Adequate organ function

Exclusion Criteria (summary):

* Patients currently participating and receiving study therapy or patients who have participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Patients with a diagnosis of immunodeficiency, patients receiving systemic steroid therapy or, patients who have received any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Patients with a known history of active Tuberculosis
* Hypersensitivity to pembrolizumab or any of its excipients
* Prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1. Patients who have not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier are excluded.
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1. Patients who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Active autoimmune disease that has required systemic treatment in the past 2 years.
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Active infection requiring systemic therapy.
* Pregnancy
* Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent within the prior 24 weeks.
* Known history of Human Immunodeficiency Virus (HIV)
* Receipt of a live vaccine within 30 days of planned start of study therapy.
* HIFU must not be applied to a breast with an implant. A region outside of the breast may be targeted as long as the targeted area is at least 10mm away from an implant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Dillon, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Sheybani ND, Witter AR, Thim EA, Yagita H, Bullock TNJ, Price RJ. Combination of thermally ablative focused ultrasound with gemcitabine controls breast cancer via adaptive immunity. J Immunother Cancer. 2020 Aug;8(2):e001008. doi: 10.1136/jitc-2020-001008. PMID 32819975

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: 1st Dose of Pembrolizumab After HIFU | Arm B: 1st Dose of Pembrolizumab Before HIFU
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: 1st Dose of Pembrolizumab After HIFU | Arm B: 1st Dose of Pembrolizumab Before HIFU | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Customized [Mean (Standard Deviation); unit: years] | 47.7 (10.3) | 57.9 (9.63) | 53.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 7 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 3 | 4 | 7
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 13
Eastern Cooperative Oncology Group (ECOG) Performance Status [Mean (Full Range); unit: units on a scale] — 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead Numeric values that are lower indicate "better"
  units on a scale | 1.2 [0 to 2] | 1.3 [0 to 2] | 1.2 [0 to 2]

OUTCOME MEASURES:

1. Primary Outcome: Change in Proportion of CD8+ Tumor Infiltrating Lymphocytes
Description: How many of the immune cells inside a tumor are a specific type of "killer" T cell
Time Frame: baseline and week 4
Population: The ratio of CD8/CD4 in the periablated zone around the tumor is described as mean of the ratios of CD8/CD4 in each patient collected by ultrasound guided needle biopsy in the peri-ablated tumor area (within 10mm of ablation margin)
Measure: Mean (Standard Deviation); unit: ratio of CD8 to CD4
Arm/Group | Arm A: 1st Dose of Pembrolizumab After HIFU | Arm B: 1st Dose of Pembrolizumab Before HIFU
Number analyzed (Participants) | 6 | 7
ratio of CD8 to CD4 | 35.98 (64.38) | 126.39 (216.16)

ADVERSE EVENTS:
Time Frame: AEs were collected from the time treatment begins until end of treatment (about 1 year).
Arm/Group | Arm A: 1st Dose of Pembrolizumab After HIFU | Arm B: 1st Dose of Pembrolizumab Before HIFU
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/6 | 3/7
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: 1st Dose of Pembrolizumab After HIFU (N=6) | Arm B: 1st Dose of Pembrolizumab Before HIFU (N=7)
Blood Bilirubin Increased (Investigations) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Alkaline Phosphatase Increased (Investigations) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: 1st Dose of Pembrolizumab After HIFU (N=6) | Arm B: 1st Dose of Pembrolizumab Before HIFU (N=7)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 3 (3)
Pain (General disorders) | 2 (2) | 1 (1)
Bruising (General disorders) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Weight Loss (Investigations) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
The study terminated early due to difficulty with enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/72/NCT03237572/Prot_SAP_001.pdf
  • Informed Consent Form (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT03237572/ICF_000.pdf